CLINICAL TRIAL: NCT02095093
Title: Intellijoint HIP Limited Release Trial: An Intelligent Instrument for Improved Leg Length and Hip Offset Accuracy in Total Hip Arthroplasty
Brief Title: An Intelligent Instrument for Improved Leg Length and Hip Offset Accuracy in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Intellijoint HIP
Record Dates: First submitted 2013-11-08; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Hip Osteoarthritis; Leg Length Discrepancy; Dislocation
Keywords: Total Hip Arthroplasty; Navigation; Imageless; THA; Computer navigated
MeSH Terms: conditions — Osteoarthritis, Hip; Leg Length Inequality; Joint Dislocations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intellijoint HIP (Experimental): Patient's will have their leg length and hip offset determined intraoperatively using Intellijoint HIP.
  Interventions: Device: Intellijoint HIP
- Outrigger (Active Comparator): Control patients will have their leg length and hip offset determined intra-operatively using the standard at Mount Sinai Hospital, which is a pin and outrigger system.
  Interventions: Device: Outrigger

INTERVENTIONS:
Device: Intellijoint HIP — Intellijoint HIP is an intra-operative, imageless intelligent instrument used to provide real-time information to surgeons about leg length and hip offset changes during total hip replacement surgery.
  Arms: Intellijoint HIP
Device: Outrigger — The outrigger is a pin and caliper device that is used to assess leg length and offset during total hip arthroplasty. It is the current standard of care at Mount Sinai Hospital.
  Arms: Outrigger

SUMMARY:
Leg length discrepancies following total hip arthroplasty have been associated with nerve palsies, gait abnormalities, and lower back pain. Leg length discrepancies are related to poorer functional outcomes and patient dissatisfaction. Failure to restore femoral offset following total hip arthroplasty has been linked to decreased range of motion and abductor muscle strength, impingement, limping, higher dislocation rates, increased polyethylene wear, and loosening of implants. Computer navigation has shown to improve the accuracy of leg length and hip offset during total hip arthroplasty. The investigators research objective is to prove the accuracy of the Intellijoint HIP™ system for determining leg length and hip offset. The investigators hypothesis was that Intellijoint HIP™, an imageless intraoperative intelligent instrument, could improve the accuracy of leg length and hip offset during primary total hip arthroplasty. The investigators plan to study this hypothesis in humans by comparing the leg length and hip offset discrepancies produced with Intellijoint HIP™ to the standard at the investigators institution, which is a pin and outrigger system.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is undergoing a primary total hip arthroplasty at Mount Sinai Hospital.

Exclusion Criteria:

* Pre-operative flexion contracture >30°, infection, or inability to achieve rigid fixation of instruments intra-operatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of leg length | 6 weeks post-op
  Standard post-operative anteroposterior pelvis radiographs will be used to assess the leg length discrepancy
Accuracy of Hip Offset | 6 weeks post-op
  Standard post-operative anteroposterior pelvis radiographs will be used to assess the hip offset restoration

SECONDARY OUTCOMES:
Time of surgery | Measured at the time of surgery
  We will measure the skin-to-closure time for each surgery to assess additional time, if any, added to procedure when using PelvAssist.
Harris Hip Score | 1 year
  We will measure the Harris Hip Scores at 6 weeks and 1 year post-op.
Dislocation Rates | 1 Year
  We will record the dislocation rates at one year following surgery.
Oxford Hip Scores | 6 weeks and 1 year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kuzyk, MD, Principal Investigator — Mount Sinai Hospital, Division of Orthopedic Surgery
Locations (1):
- Mount Sinai Hospital, Torono, Ontario, Canada